CLINICAL TRIAL: NCT02405039
Title: A Multi-Center, Double-Masked, Randomized, One-Year Safety Study of EBI-005 5 mg/mL Topical Ophthalmic Solution Versus Vehicle-Control in Subjects With Dry Eye Disease (DED)
Brief Title: Study of EBI-005 in Dry Eye Disease (DED)
Acronym: EBI-005
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eleven Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: EBI-005-4
Record Dates: First submitted 2015-01-06; First posted 2015-04-01 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Dry Eye
Keywords: DED; Disease
MeSH Terms: conditions — Dry Eye Syndromes; Disease | interventions — EBI-005

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator: EBI-005 (Active Comparator): Drug: EBI-005 The investigational drug EBI-005, is an intervention to one of two study arms: 5 mg/mL topical administered 3 times per day
  Interventions: Drug: EBI-005
- Placebo or Vehicle control Comparator (Placebo Comparator): One of two study arms: placebo or vehicle control topical administered 3 times per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EBI-005 — EBI-005 is an intervention into one of two (2) study arms; 5 mg/mL topical administered 3 times per day
  Arms: Active Comparator: EBI-005
Drug: Placebo — Placebo or Vehicle control comparator is an intervention into one of two (2) study arms; vehicle topical administered 3 times per day
  Arms: Placebo or Vehicle control Comparator

SUMMARY:
This is a randomized, double masked study designed to evaluate the safety of EBI-005 5 mg/mL topical ophthalmic solution given three times daily (TID) compared to vehicle-control over a one year period in subjects with dry eye disease (DED). Approximately 188 subjects will be enrolled to either EBI-005 or vehicle at up to 15 centers in the United States (US) and Canada.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have a history of dry eye disease (DED) in both eyes supported by a previous clinical diagnosis or have a self-reported history of subjective complaints for at least 6 months prior to Visit 1
2. Are willing and able to follow instructions and can be present for the required study visits for the duration of the study

Key Exclusion Criteria:

1. Have an ocular condition that could confound study assessments (ocular infection, herpetic or neurotrophic keratitis, Steven-Johnson Syndrome, etc)
2. Have had penetrating intraocular surgery within 12 months prior to Visit 1
3. Be unwilling to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Safety of EBI-005 (vital signs) | 1 year
  Safety will be assessed by vital signs, laboratory changes over time, adverse events, and assessment of antibody development (immunogenicity) over time.
tolerability of EBI-005 (adverse events) | 1 year
  Safety will be assessed by vital signs, laboratory changes over time, adverse events, and assessment of antibody development (immunogenicity) over time.
Immunogenicity of EBI-005 (assessment of antibody development (immunogenicity) over time) | 1 year
  Safety will be assessed by vital signs, laboratory changes over time, adverse events, and assessment of antibody development (immunogenicity) over time.
Safety of EBI-005 (laboratory changes over time) | 1 year

SECONDARY OUTCOMES:
Biological effect of EBI-005 (Changes over time in the OSDI) | 1 year
  Changes over time in the OSDI.
Biological effect of EBI-005 (Total corneal fluorescein staining) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldstein, MD, Study Director — Eleven Biotherapeutics
Locations (12):
- United States (12):
  - Birmingham, Alabama
  - Newport Beach, California
  - Hamden, Connecticut
  - New Albany, Indiana
  - Louisville, Kentucky
  - Winchester, Massachusetts
  - St Louis, Missouri
  - Asheville, North Carolina
  - Mason, Ohio
  - Cranberry Township, Pennsylvania
  - Memphis, Tennessee
  - San Antonio, Texas